CLINICAL TRIAL: NCT03888001
Title: The Efficacy of Botulinum Toxin in OVERACTIVE Bladder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, AHMED FARAHAT HASSAN, principle invistigator, Assiut University
Other Study IDs: Botox in overactive bladder
Record Dates: First submitted 2019-03-18; First posted 2019-03-25 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To assess the efficacy of botulinum toxin injection in overactive bladder.

DETAILED DESCRIPTION:
Detrusor overactivity is defined as a urodynamic observation characterized by involuntary detrusor contractions during the filling phase that may be spontaneous or provoked. Detrusor overactivity is subdivided into idiopathic detrusor overactivity and neurogenic detrusor overactivity The International Continence Society (ICS) defines OAB as the presence of "urinary urgency, usually accompanied by frequency and nocturia, with or without urgency urinary incontinence, in the absence of UTI or other obvious pathology. Neurogenic detrusor overactivity (NDO) can result in lower and upper urinary tract complications and eventually even in end-stage kidney failure. Since the driving force of this clinical cascade is high bladder pressure, controlling intravesical pressure in NDO patients improves both quality of life and life-expectancy in these patients. Botulinum toxin A (BTX-A) has proven its efficacy in reducing intravesical pressure and in reducing incontinence episodes. BTX-A also improves quality of life in patients with NDO. Both onabotulinumtoxinA (Botox®, Allergan, Irvine, USA) and abobotulinumtoxinA (Dysport®, Ipsen, Paris, France) have a level A recommendation for NDO-treatment. The recommended dose for intradetrusor injections in NDO patients is 200 U of onabotulinumtoxinA or 500 U of abobotulinumtoxinA. The drug is generally administered extratrigonal in the detrusor muscle, via cystoscopic guided injection at 20 sites in 1 mL injections. Intradetrusor BTX-A injections are safe, with mostly local complications such as urinary tract infection and high post-void residual or retention. The effect of the toxin lasts for approximately 9 months. Repeat injections can be performed without loss of efficacy. Different injection techniques, novel ways of BTX-A administration, eliminating the need for injection or new BTX-A types with better/longer response rates could change the field in the future. Botulinum toxins are neurotoxins produced by the facultative anaerobe Clostridium botulinum that block the release of acetylcholine into the synaptic gap of the neuromuscular junction. Their injection near the nerves that supply the target organ selectively and temporarily paralyzes the organ. In particular, the subtype botulinum-A toxin is widely used in neurology to release spastic dystonia in adults. and children. In urologic disorders, botulinum-A toxin reliably diminishes external sphincter or detrusor overactivity.

ELIGIBILITY:
1. Inclusion criteria:

   * patients with spastic neurogenic bladder due to upper motor neuron lesion as (spinal cord lesions ,multiple sclerosis ,strokes,parkinsonism...........).
   * patients with idiopathic overactive bladder
   * patients with spastic neurogenic bladder diagnosed clinically and urodynamically.
2. Exclusion criteria:

   * patients with diabetes mellitus.
   * Atonic bladder.
   * Children below 6 years.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with either sex and above age of 6 years with diagnosis of idiopathic or neurogenic overactive bladder diagnosed clinically and urodynamically admitted to Assiut university hospital. Paitent with neurogenic lowcompliance or detrusor overactivity affecting bladder function
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-04-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Botulinum Toxin injection in overactive Bladder | 1 year
  By using of quistionaire mainly arabic validation of urogenital distress inventory ( UDI-6 quistionaire) throug appling quistions to patients that compare between symptoms before and after botox injection...

CONTACTS AND LOCATIONS:
Overall Officials: AHMED FARAHAT, MASTER, Principal Investigator — Assiut University
Locations (1):
- Ahmed Farahat, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1. Fowler CJ, Griffiths D, de Groat WC. The neural control of micturition. Nat Rev Neurosci 2008;9:453-66. 2. Aoki KR, Guyer B. Botulinum toxin type A and other botulinum toxin serotypes: a comparative review of biochemical and pharmacological actions. Eur J Neurol 2001;8 Suppl 5:21-9. 3. Tanagho EA, McAninch JW, editors. Smith's General Urology. 17th ed. New York: The McGraw-Hill Companies, Inc., 2008,438-53. 4. Sellers DJ, McKay N. Developments in the pharmacotherapy of the overactive bladder. Curr Opin Urol2007;17:223-30. 5-Aoki, K.R. Pharmacology and immunology of botulinum toxin serotypes. J. Neurol. 2001; 248: 3-10